CLINICAL TRIAL: NCT00651911
Title: A Multicenter Open Label Study of the Efficacy and Safety of Rasburicase in the Treatment of Prophylysis for Tumor Lysis Syndrome
Brief Title: Fasturtec TLS Treatment / Prophylysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8637
Record Dates: First submitted 2008-03-28; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Tumor Lysis Syndrome
MeSH Terms: conditions — Tumor Lysis Syndrome | interventions — Urate Oxidase; rasburicase

INTERVENTIONS:
Drug: urate oxidase — First injection of Rasburicase will be done the day of initiation of chemotherapy, or the day before, according to hyperuricemia. Additional doses are permitted q12h during the first 72 hours of chemotherapy if hyperuricemia persists or subject is considered to be at significant risk of tumor lysis complications.
  Other Names: rasburicase

SUMMARY:
An open-label study to determine the efficacy and safety of Rasburicase used for the prevention and treatment of tumor lysis syndrome

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy planned for at least 3 cycles
* Undergoing cytoreductive chemotherapy for ALL, multiple myeloma or Burkitt's lymphoma stage III or IV
* With a minimum life expectancy of 3 months
* Uric acid > 8 mg%
* Negative pregnancy test < or =to 2 weeks and efficient contraceptive method.
* Negative HIV serology < or =to 4 weeks
* Patient or legal guardian has signed a written informed consent

Exclusion Criteria:

* Hypersensitivity to uricases or any of the excipients
* Known history of G6PD deficiency.
* Previous treatment with Rasburicase or Uricozyme®
* Pregnancy or lactation
* Treatment with any investigational drug within 30 days before planned first Rasburicase administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-07; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
To assess the uricolytic response to rasburicase treatment | 5 weeks (3 to 7 days of treatment, with follow-up of 4 weeks after the last study drug injection)

SECONDARY OUTCOMES:
To evaluate tumor lysis risk factors, treatments for tumor lysis syndrome and complications of treatment in patients treated prophylactically or therapeutically for tumor lysis syndrome | 5 weeks (3 to 7 days of treatment, with follow-up of 4 weeks after the last study drug injection)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chang, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States